CLINICAL TRIAL: NCT01190865
Title: A Phase I Study Investigating the Survival of HP802-247 Allogeneic Cells in Excisional Acute Cutaneous Wounds
Brief Title: Study of Survival Duration for Donor Skin Cells in Skin Biopsy Wounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802-247-09-021
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Normal Female Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HP802-247 (Other): Assessment Duration = 8 days Assessment Duration = 15 days Assessment Duration = 22 days Assessment Duration = 29 days Assessment Duration = 31 days Assessment Duration = 43 days Assessment Duration = 50 days Assessment Duration = 57 days
  Interventions: Biological: HP802-247

INTERVENTIONS:
Biological: HP802-247 — One dose of HP802-247 consisting off 260 mL containing keratinocytes and fibroblasts totaling 5.0 x 10.6 cells per mL, plus fibrin.

SUMMARY:
The goal for this study is to examine the persistence of growth arrested,allogeneic,male-donor keratinocytes and fibroblasts when applied as product HP802-247 to the surface of acute excisional wounds in health female volunteers, as measured using Y-STR for detection of Y-chromosome.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Female, 18 years of age or older.
* Any race or skin type, provided that there are no tattoos within 5 cm of the wound target, and the gentian violet surgical marker produces a clearly visible mark on the skin.
* Willing to make all required study visits and, in the opinion of the Investigator, able to follow instructions.
* Willing to undergo the repeated biopsy procedures.
* Willing to undergo verification of sex chromosome status.

Exclusion Criteria:

* Males, or phenotypic females bearing Y-chromosome genetic material [e.g., 46,X,(r)Y; 46,X,der(X)t(X;Y); sex reassignment surgery].
* Contraindications or hypersensitivity to the use of the study medications or their components (e.g., history of anaphylaxis, serum sickness, or erythema multiforme reaction to aprotinin, bovine serum albumin or bovine serum proteins, penicillin, streptomycin, or amphotericin B).
* History of keloid formation or hypertrophic scarring.
* Participation in any interventional clinical trial within 30 days prior to screening.
* History of prolonged bleeding, bleeding into joints, easy bruising following minor trauma, clotting factor deficiency, or current use of anticoagulants or platelet inhibitors.
* Any medical condition which, in the opinion of the Co-Investigator, may interfere with normal wound repair.
* Current therapy with drugs or biologics intended to function as immuno-suppressants, chronic (> 10 days) oral corticosteroids, or any concomitant medication which, in the opinion of the Co-Investigator, may interfere with normal wound repair.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint, Ltd; Barry Reece, MS, Principal Investigator — RCTS, Inc.
Locations (1):
- RCTS, Inc., Irving, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a single US investigational site, between September 14, 2010 and December 08, 2010.
Pre-assignment Details: Subjects underwent buccal smear to ensure absence of a Y chromosome or translocated material from a Y chromosome. Day 1, all subjects underwent a baseline 3mm skin punch biopsy on the inner upper arm followed by a single application of HP802-247.
Period: Overall Study
Arm/Group | HP802-247
Started | 28
Completed | 25
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | HP802-247
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Identification of the Full Set of Y-chromosome Short Tandem Repeats in Each Bioopsy.
Description: The primary efficacy variable was detection of the full set of 17 Y STR loci. If all loci amplified such that a clear identification of a donor was possible, the test result was categorized as positive. If fewer loci amplified such that identification of the donor was not possible in a forensic setting, the result was categorized as negative. Descriptive statistics are presented for this variable.
Time Frame: Cohorts of 3 subjects were biopsied at weekly intervals for 8 weeks
Population: 3 subjects were withdrawn; 2 for non-compliance and one at the subject's request. One subject, who was available to replace a subject assigned to a weekly cohort if the subject was unavailable, was assayed on Day 57 with the subjects assigned to the Week 8 cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | HP802-247
Number analyzed (Participants) | 25
Participants
  Week 1, Day 8: number analyzed (Participants) | 3
  Week 1, Day 8 | 3
  Week 2, Day 15: number analyzed (Participants) | 3
  Week 2, Day 15 | 1
  Week 3, Day 22: number analyzed (Participants) | 3
  Week 3, Day 22 | 0
  Week 4, Day 29: number analyzed (Participants) | 3
  Week 4, Day 29 | 0
  Week 5, Day 36: number analyzed (Participants) | 3
  Week 5, Day 36 | 0
  Week 6, Day 43: number analyzed (Participants) | 3
  Week 6, Day 43 | 0
  Week 7, Day 50: number analyzed (Participants) | 3
  Week 7, Day 50 | 0
  Week 8 Day 57: number analyzed (Participants) | 4
  Week 8 Day 57 | 0

2. Secondary Outcome: Time in Days to 50% Correct Identification (ID50) of the Implanted Male DNA 17 Loci in Female Volunteers, With Regard to Three DNA Profile Types, Including Partial DNA Profile, > 50% DNA Profile, and Full (or Complete) DNA Profile.
Description: The biopsy area was examined for the presence of the Y chromosome, based on the presence of a full set of Y-STR loci as well as partial sets, assayed by a commercial kit (AmpFISTRTM).
  Probit analysis was utilized to determine the time in days to 50% correct identification (ID50) of the implanted male DNA 17 loci in female volunteers, with regard to three DNA profile types, including partial DNA profile, > 50% DNA profile, and full (or complete) DNA profile. The analysis was performed using SAS® PROC PROBIT
Time Frame: Cohorts of 3 subjects were biopsied at weekly intervals for 8 weeks
Population: The analysis population consisted of the 8 cohorts of 3 subjects biopsied at weekly intervals over the 8-week duration of the study. It should be note that the cohort for Week 8 (Day 57) was composed of 4 subjects
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | HP802-247
Number analyzed (Participants) | 25
Days
  Partial DNA profile | 19 [0 to 30]
  ≥ 50% of the 17 loci | 17 [0 to 28]
  Complete DNA profile | 13 [0 to 24]

ADVERSE EVENTS:
Time Frame: Safety reporting occurred over the eight weeks of the study.
Description: All subjects randomized to treatment were questioned about adverse events and were included in the number of participants assessed for safety. The first assessments at each visit were about changes in general health and concomitant medications and the occurrence of adverse events.
Arm/Group | HP802-247
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 8/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=28)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 (N=28)
Furuncle (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Urinary Tract Infection (UTI) (Infections and infestations) | 1 (1)
Human Bite (Injury, poisoning and procedural complications) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1)
Blood Cholesterol Increase (Investigations) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less